CLINICAL TRIAL: NCT00003021
Title: A Phase I Trial of Bizelesin (NSC 615291) Using a Single Bolus Infusion Given Every Twenty-eight (28) Days in Patients With Advanced Cancer
Brief Title: Bizelesin in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065606; UTHSC-IDD-93-45; NCI-T93-0166; SACI-IDD-93-45
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — bizelesin

INTERVENTIONS:
Drug: bizelesin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of bizelesin in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of bizelesin in patients with advanced cancer. II. Determine the qualitative and quantitative toxic effects of this therapy in these patients. III. Determine the pharmacokinetics of this therapy in these patients. IV. Determine the recommended dose of this drug for phase II trials. V. Determine the antitumor effects of this therapy in these patients.

OUTLINE: This is a dose-escalation study. Patients receive bizelesin IV on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of bizelesin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant solid tumor for which there are no therapeutic options that are potentially curative or have been demonstrated to increase survival No primary or metastatic CNS malignancy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin normal SGOT no greater than 2.5 times upper limit of normal Renal: Creatinine normal OR Creatinine clearance at least 60 mL/min Cardiovascular: No atrial or ventricular arrhythmia requiring medication No ischemic event within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection No other active malignancy except curatively treated carcinoma in situ of the cervix or basal cell skin cancer No other serious concurrent medical illness No history of seizure disorder requiring active therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to more than 10% of bone marrow No prior electron-beam radiotherapy At least 4 weeks since other prior radiotherapy Surgery: Prior surgery allowed Other: Recovered from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-08; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas